CLINICAL TRIAL: NCT02973724
Title: Predicted EC95 of Effect-site Concentration of Remifentanil for Preventing Cough After Laryngomicrosurgery From Propofol Anesthesia
Brief Title: EC95 of Remifentanil for Preventing Cough
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jong Yeop Kim, Professor, Ajou University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AJIRB-MED-CT4-16-349
Record Dates: First submitted 2016-11-21; First posted 2016-11-25 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Drug Usage
Keywords: Extubation; Remifentanil; Laryngomicrosurgery
MeSH Terms: interventions — Remifentanil; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Remifentanil (Experimental): Extubation was performed when remifentanil was maintained a predetermined concentration throughout the emergence periods.
  Interventions: Drug: Remifentanil; Drug: Propofol anesthesia

INTERVENTIONS:
Drug: Remifentanil — The concentration of remifentanil was determined by biased-coin up and down design, starting from 1.0 ng/ml (0.4 ng/ml as a step size)
  Other Names: Ultiva
Drug: Propofol anesthesia — Anesthesia was induced with propofol target-controlled infusion at an effect-site concentration of 5.0 μg/ml.
  Other Names: Fresofol

SUMMARY:
The investigator designed this study to investigate remifentanil effect-site concentration in 95% of patients (EC95) for preventing cough after laryngomicrosurgery from propofol anesthesia.

DETAILED DESCRIPTION:
At the end of the surgery, propofol infusion was stopped and remifentanil was titrated to predetermined (initial concentration 1.0 ng/ml for the first patient). Extubation was performed when the patients opened their eyes and spontaneous respiration and adequate tidal volume and ventilatory frequency were confirmed.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II patients undergoing general anesthesia for laryngomicrosurgery

Exclusion Criteria:

* Anticipated difficult airway
* COPD, Asthma
* Recent URI (< 2 weeks)
* Severe cardiac, hepatic renal disease

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Number of cough | from end of surgery to 5 min after tracheal extubation
  Number of cough or a strong and sudden contraction of the abdomen during periextubation periods

CONTACTS AND LOCATIONS:
Locations (1):
- Ajou University Hospital, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No